CLINICAL TRIAL: NCT03172624
Title: A Phase II Study of Nivolumab Plus Ipilimumab in Patients With Recurrent/Metastatic Salivary Cancers
Brief Title: Study of Nivolumab Plus Ipilimumab in Patients With Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-219
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-12

CONDITIONS: Salivary Gland Cancer
Keywords: Nivolumab; Ipilimumab; 17-219
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: This is a phase II study evaluating the efficacy of nivolumab in combination with ipilimumab in patients with recurrent and/or metastatic (R/M) salivary gland cancers (SGCs). Patients will be enrolled to two cohorts: Cohort 1, patients with R/M adenoid cystic carcinoma ("ACC group"), and Cohort 2: patients with R/M SGC of any histology, except ACC ("non-ACC group").
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- R/M adenoid cystic carcinoma (ACC) (Experimental): Enrolled patients will be treated with nivolumab 3 mg/kg every 2 weeks plus ipilimumab 1 mg/kg every 6 weeks (1 cycle= 6 weeks).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- R/M SGC of any histology, except ACC (Non ACC) (Experimental): Enrolled patients will be treated with nivolumab 3 mg/kg every 2 weeks plus ipilimumab 1 mg/kg every 6 weeks (1 cycle= 6 weeks).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — nivolumab 3 mg/kg every 2 weeks
Drug: Ipilimumab — ipilimumab 1 mg/kg every 6 weeks (1 cycle= 6 weeks)

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, treatment with two drugs called nivolumab and ipilimumab have on the participant and salivary cancer.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 only: Patients must have pathologically or cytologically confirmed adenoid cystic carcinoma. Cancers arising from non-salivary gland primary sites are allowed.
* Patients must have pathologically or cytologically confirmed salivary gland cancer of any histology except for adenoid cystic carcinoma.
* Patients must have recurrent and/or metastatic disease not amenable to potentially curative surgery or radiotherapy.
* At least 2 weeks must have elapsed since the end of prior systemic treatment and/or 4 weeks since completion of radiotherapy with resolution of all treatment-related toxicity to NCI CTCAE Version 4.0 grade ≤1 (or tolerable grade 2) or back to baseline (except for alopecia, lymphopenia, or hypothyroidism) prior to starting study drug treatment. Any number of prior therapies for recurrent/metastatic salivary gland cancer are allowed.

NOTE: Patients previously treated with hormonal therapies (e.g., drugs targeting the androgen receptor) may continue these drugs prior to trials enrollment and concomitantly with study therapy.

* Patients must have RECIST v1.1 measurable disease.
* Cohort 1 and acinic cell carcinoma patients in Cohort 2 only: Patients must have documentation of a new or progressive lesion on a radiologic imaging study performed within 6 months prior to study enrollment (progression of disease over any interval is allowed) and/or new/worsening disease related symptoms within 6 months prior to study enrollment. Note: This assessment will be performed by the treating investigator. Evidence of progression by RECIST criteria is not required.
* Age ≥ 18 years.
* ECOG performance status 0 or 1 (or Karnofsky ≥ 70%).
* Patients must have tissue from the primary tumor or metastases available for correlative studies. Either a paraffin block or at least 20 unstained slides are acceptable (30 unstained slides would be ideal). (If less than twenty unstained slides are available and a paraffin bloc is not available, the patient may be able to participate at the discretion of the investigator.)
* Patients must agree to undergo two research biopsies of malignant lesions. Tumor tissue obtained prior to study consent or treatment as part of standard of care can also be submitted in lieu of performance of the first pre-treatment biopsy, if the Principal Investigator deems it to be of sufficient quantity/quality/timeliness. Patients may be exempt from biopsy if 1) the investigator or person performing the biopsy judges that no tumor is accessible for biopsy, 2) the investigator or person performing the biopsy feels that the biopsy poses too great of a risk to the patient, or 3) the patient's platelet count is <100,000/mcl or he/she cannot be safely removed from anti-coagulation therapy (if the anti-coagulation therapy needs to be temporarily held for the biopsy procedure). If the only tumor accessible for biopsy is also the only lesion that can be used for RECIST v1.1 response evaluation, then the patient may be exempt from biopsy. If the investigator deems a second research biopsy to be high risk after a patient has completed the first research biopsy, the patient may be exempt from the second biopsy.
* Screening laboratory values must meet the following criteria:

  * WBC ≥ 2000/μL
  * Neutrophils ≥ 1500/μL
  * Platelets ≥ 100 x10^3/μL
  * Hemoglobin > 9.0 g/dL
  * AST/ALT ≤ 3 x ULN
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL

Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

* Women of childbearing potential (WOCBP)* must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.

  * WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes.

Women who are not of childbearing potential are not required to use contraception.

* Women of childbearing potential must have a negative serum or urine pregnancy test upon study entry.
* Men who are sexually active with women of child bearing potential must use adequate contraception upon study entry until 31 weeks after the last dose of study treatment. Men who are surgically sterile or azoospermic do not require contraception.

Exclusion Criteria:

* Symptomatic metastatic brain or leptomeningeal tumors (asymptomatic or treated metastatic brain or leptomeningeal tumors are allowed).
* Current or prior use of immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalents) or other immunosuppressive medications within 2 weeks of study drug administration. NOTE: Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if >10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Active, known, or suspected autoimmune disease within the past 2 years. NOTE: Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have had prior systemic treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* Patients should be excluded if they have a known history of testing positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus antibody (HCV antibody) indicating acute or chronic infection (those with treated hepatitis B or C infection and a negative viral load prior to study entry would be eligible)
* Patients should be excluded if they have a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* History of allergy to study drug components.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vos JL, Burman B, Jain S, Fitzgerald CWR, Sherman EJ, Dunn LA, Fetten JV, Michel LS, Kriplani A, Ng KK, Eng J, Tchekmedyian V, Haque S, Katabi N, Kuo F, Han CY, Nadeem Z, Yang W, Makarov V, Srivastava RM, Ostrovnaya I, Prasad M, Zuur CL, Riaz N, Pfister DG, Klebanoff CA, Chan TA, Ho AL, Morris LGT. Nivolumab plus ipilimumab in advanced salivary gland cancer: a phase 2 trial. Nat Med. 2023 Dec;29(12):3077-3089. doi: 10.1038/s41591-023-02518-x. Epub 2023 Aug 24. PMID 37620627
- [Derived] Tchekmedyian V. Salivary Gland Cancers. Hematol Oncol Clin North Am. 2021 Oct;35(5):973-990. doi: 10.1016/j.hoc.2021.05.011. PMID 34503735
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R/M Adenoid Cystic Carcinoma (ACC) | R/M SGC of Any Histology, Except ACC (Non ACC)
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R/M Adenoid Cystic Carcinoma (ACC) | R/M SGC of Any Histology, Except ACC (Non ACC) | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Median (Full Range); unit: years] | 58 [30 to 88] | 64 [57 to 88] | 64 [30 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 13 | 20 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 30 | 29 | 59
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 28 | 26 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | R/M Adenoid Cystic Carcinoma (ACC) | R/M SGC of Any Histology, Except ACC (Non ACC)
Number analyzed (Participants) | 32 | 32
Participants
  Partial Response | 2 | 5
  Stable Disease | 17 | 8
  Progressive Disease | 13 | 18
  Not Evaluable | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | R/M Adenoid Cystic Carcinoma (ACC) | R/M SGC of Any Histology, Except ACC (Non ACC)
All-Cause Mortality (participants affected / at risk) | 6/32 | 7/32
Serious Adverse Events (participants affected / at risk) | 18/32 | 9/32
Other Adverse Events (participants affected / at risk) | 11/32 | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R/M Adenoid Cystic Carcinoma (ACC) (N=32) | R/M SGC of Any Histology, Except ACC (Non ACC) (N=32)
Alanine aminotransferase increased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Ejection fraction decreased (Cardiac disorders) | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Fever (General disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Jejunal obstruction (Gastrointestinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Malaise (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R/M Adenoid Cystic Carcinoma (ACC) (N=32) | R/M SGC of Any Histology, Except ACC (Non ACC) (N=32)
Alanine aminotransferase increased (Investigations) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4
Hyponatremia (Metabolism and nutrition disorders) | 4 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2
Lymphocyte count decreased (Investigations) | 11 | 14
Neutrophil count decreased (Investigations) | 2 | 3
White blood cell decreased (Investigations) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT03172624/Prot_SAP_000.pdf